CLINICAL TRIAL: NCT04163263
Title: Phase 1, Randomized, Vehicle-Controlled, Double-Blind Study to Evaluate the Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Effects of Repeat Topical Application of BOS-356 in Subjects With Moderate to Severe Acne Vulgaris
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Effects of Repeat Topical Application of BOS-356 in Subjects With Moderate to Severe Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: BOS-356-101
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Moderate to Severe Acne Vulgaris
Keywords: BOS-356; acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohorts 1-3: BOS-356 (Experimental): Twice daily application of BOS-356 0.1%, 0.4%, and 0.7% gel in Cohorts 1, 2, and 3, respectively
  Interventions: Drug: BOS-356
- Cohorts 1-3: Vehicle (Placebo Comparator): Twice daily application of vehicle gel
  Interventions: Drug: Vehicle
- Cohort 4: BOS-356 (Experimental): Twice daily application of BOS-356 gel at a dose determined based on safety and tolerability data from Cohorts 1-3
  Interventions: Drug: BOS-356
- Cohort 4: Vehicle (Placebo Comparator): Twice daily application of vehicle gel
  Interventions: Drug: Vehicle
- Cohort 5: BOS-356 (Experimental): Twice daily application of BOS-356 gel at a dose determined based on safety and tolerability data from Cohorts 1-3
  Interventions: Drug: BOS-356
- Cohort 5: Vehicle (Placebo Comparator): Twice daily application of vehicle gel
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: BOS-356 — topical gel
  Arms: Cohort 4: BOS-356; Cohort 5: BOS-356; Cohorts 1-3: BOS-356
Drug: Vehicle — topical gel
  Arms: Cohort 4: Vehicle; Cohort 5: Vehicle; Cohorts 1-3: Vehicle

SUMMARY:
This study is being conducted to characterize the safety and tolerability of BOS-356 in adult participants with moderate to severe acne vulgaris following 14 days or 28 days of repeated topical application

DETAILED DESCRIPTION:
In Cohorts 1-3, participants will be randomized to receive twice daily (BID) topical applications of BOS-356 gel or vehicle gel to the face during a 14-day treatment period. Doses will be escalated in successive cohorts with BOS-356 gel 0.1%, 0.4%, and 0.7%.

In Cohort 4, participants will be randomized to receive BID topical applications of BOS-356 gel or vehicle gel to the face, upper chest, upper back, shoulders, and posterior neck during a 28-day treatment period. The dose of BOS-356 to be used in this cohort will be determined based on safety and tolerability data from Cohorts 1-3.

In Cohort 5, participants will complete a 7-day run-in period to receive BID topical applications of vehicle gel to the face. Participants will be randomized to receive BID topical applications of BOS-356 gel or vehicle gel to the face during a 28-day treatment period. The dose of BOS-356 to be used in this cohort will be the same as the dose used in Cohort 4. Cohorts 4 and 5 may proceed in parallel.

ELIGIBILITY:
Inclusion Criteria:

For Cohorts 1-5:

* Male or female participants aged 18 to 45 years, inclusive, at the time of consent
* Participant has moderate to severe non-nodular facial acne vulgaris.
* Participant's treatment with hormonal therapy (including, but not limited to, topical application, oral administration, implant, intrauterine device [IUD]) has been on a stable dose and frequency for at least 12 weeks before Day 1, and participant agrees to maintain current dose and frequency throughout the study.
* Female participants of childbearing potential and male participants and their female partners who are of childbearing potential must agree to use a highly effective contraceptive method
* Participant is willing to participate and is capable of giving informed consent. Note: Consent must be obtained prior to any study-related procedures.

Additional Inclusion Criteria for Cohort 4 only:

• Participant has additional acne lesions on the upper back with at least 5 inflammatory lesions and additional acne lesions on the posterior neck, shoulders, and/or upper chest.

Exclusion Criteria:

For Cohorts 1-5:

* Participant is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
* Participant has acne fulminans, conglobata, nodulocystic acne, or secondary acne.
* Participant has a history of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the study assessments.
* Excessive facial hair that would interfere with diagnosis or assessment of acne vulgaris
* Participant is known to have immune deficiency or is immunocompromised.
* Participant has a history of cancer or lymphoproliferative disease within 5 years prior to Day 1. Participants with successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix may be candidates for the study.
* Participant had a major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study.
* Participant has positive results for hepatitis B surface antigens (HBsAg), antibodies to hepatitis B core antigens (anti-HBc), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
* Participant has used on the treated areas an over-the-counter (OTC) topical medication for the treatment of acne vulgaris, including benzoyl peroxide, topical anti-inflammatory medications, corticosteroids, salicylic acid, α-hydroxy/glycolic, or antibacterial/antiseptic soap or wash within 2 weeks prior to Day 1.
* Participant has used prescription topical retinoid (e.g., tretinoin, tazarotene, adapalene), dapsone or antimicrobials (e.g., clindamycin, erythromycin), or other prescription topical medications for the treatment of acne vulgaris within 4 weeks prior to Day 1. Topical antibiotics may be used to treat non-acne skin lesions outside of the treated area.
* Participant has used systemic antibiotics or other systemic anti-acne drugs not mentioned in other exclusion criteria within 4 weeks prior to Day 1.
* Participant has used oral or injectable corticosteroids within 4 weeks prior to Day 1 or require them during the study. Note: Intranasal corticosteroids and inhaled corticosteroids are allowed. Eye and ear drops containing corticosteroids are also allowed.
* Participant had a facial procedure (including, but not limited to, chemical peel, laser, microdermabrasion) within 8 weeks prior to Day 1 and during the study.
* Participant has received photodynamic therapy or phototherapy within 12 weeks of Day 1.
* Participant has used androgen receptor blockers (such as spironolactone or flutamide) within 12 weeks prior to Day 1.
* Participant has used drospirenone, chlormadinone acetate, or cyproterone acetate within 26 weeks prior to Day 1.
* Participant has used oral retinoid (e.g., isotretinoin) within 52 weeks prior to Day 1 or vitamin A supplements >10,000 Units per day (U/d) within 26 weeks prior to Day 1.
* Participant is currently receiving a nonbiological investigational product or device or has received one within 4 weeks or five half-lives (whichever is longer) prior to Day 1.
* Participant has received blue light, laser, intense pulsed light or other light therapy on the face within 4 weeks prior to Day 1.
* Participants who have given > 50 milliliters (mL) of blood or plasma within 30 days of Screening or > 499 mL of blood or plasma within 56 days of Screening (during a clinical trial or at a blood bank donation).
* Participant has a known history of clinically significant drug or alcohol abuse in the last year prior to Day 1, or has a positive drug screen and/or positive alcohol test result at the Screening visit or at Day 1 (excluding cannabinoids).
* Participant has had excessive sun exposure or has used tanning booths within 4 weeks prior to Day 1 or is not willing to minimize natural and artificial sunlight exposure during the study. Use of sunscreen products (except on treated areas) and protective apparel are recommended when sun exposure cannot be avoided.

For Cohorts 1-3 only:

• Participant has a Fitzpatrick's Skin Phototype ≥5.

For Cohort 4 only, due to biopsy collection:

* Participant has a history of an allergic reaction or significant sensitivity to lidocaine or other local anesthetics.
* Participant has a history of hypertrophic scarring or keloid.
* Participant has taken anticoagulant medication, such as heparin, low molecular weight (LMW)-heparin, warfarin, antiplatelets, within 2 weeks prior to Day 1, or has a contraindication to skin biopsies. Nonsteroidal anti-inflammatory drugs (NSAIDs) will not be considered antiplatelets and will be allowed.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Cohorts 1-3: Number of participants with any adverse event (AE) and any serious adverse event (SAE) | up to Day 21 for each cohort
Cohorts 1-3: Number of participants with a mild, moderate, and severe score in local tolerability assessments (LTAs) | up to Day 21 for each cohort
Cohorts 1-3: Number of participants with any clinically significant change from baseline in clinical laboratory parameter values | up to Day 21 for each cohort
Cohorts 1-3: Number of participants with any clinically significant change from baseline in vital sign values | up to Day 21 for each cohort
Cohorts 1-3: Number of participants with any clinically significant change from baseline in electrocardiogram (ECG) findings | up to Day 14 for each cohort
Cohort 4: Number of participants with any AE and any SAE | up to Day 35
Cohort 5: Number of participants with any AE and any SAE | up to Day 42
Cohort 4: Number of participants with a mild, moderate, and severe score in LTAs | up to Day 35
Cohort 5: Number of participants with a mild, moderate, and severe score in LTAs | up to Day 42
Cohorts 4 and 5: Number of participants with any clinically significant change from baseline in clinical laboratory parameter values | up to Day 35 for each cohort
Cohorts 4 and 5: Number of participants with any clinically significant change from baseline in vital sign values | up to Day 35 for each cohort
Cohorts 4 and 5: Number of participants with any clinically significant change from baseline in ECG findings | up to Day 35 for each cohort

SECONDARY OUTCOMES:
Cohorts 1-3: Plasma concentration of BOS-356 | up to Day 21 for each cohort
  Days 1 and 14: pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours post morning (AM) dose. Days 2 and 7: pre-dose; 1 and 2 hours post AM dose. Day 15: 24 hours (± 2 hours) post last dose. Follow-Up visit (Day 21) (or end-of-treatment, if applicable): at time of visit
Cohort 4: Plasma concentration of BOS-356 | up to Day 35
  Days 1 and 14: pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours post AM dose. Days 2, 7, and 15: pre-dose; 1 and 2 hours post AM dose. Day 28: pre-dose; 1, 2, 4, 6, and 8 hours post AM dose. Follow-Up visit (Day 35) (or end-of-treatment, if applicable): at time of visit
Cohort 5: Plasma concentration of BOS-356 | up to Day 35
  Day 1: pre-dose. Days 7, 14, and 28 pre-dose (approximately 12 hours [± 4 hours] from the previous dose. Follow-Up visit (Day 35): at time of visit

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Center for Dermatology Clinical Research, Fremont, California
  - International Clinical Research, Sanford, Florida
  - Dermatology Consulting Services, High Point, North Carolina
  - DermResearch, Inc., Austin, Texas
  - J&S Studies, Inc., College Station, Texas
  - Progressive Clinical Research, San Antonio, Texas
- Innovaderm Research, Inc., Montreal, Canada

IPD SHARING:
Plan to Share IPD: No